CLINICAL TRIAL: NCT06548659
Title: The Effect Of Screen-Based Sımulatıon Traınıng On Self-Effıcacy In Pedıatrıc Drug Applıcatıons And Self-Confıdence In Learnıng Among Nursıng Students
Brief Title: The Effect of Screen-Based Simulation Training on Self-Efficacy and Self-Confidence in Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Hilal Çelik Bayram, Nurse Practitioner, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0000-0003-1659-3464
Record Dates: First submitted 2024-07-17; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Educational Problems
Keywords: Nursing education; simulation

STUDY DESIGN:
Intervention Model Description: Randomization took place among 198 people. While the intervention group was given training on pediatric medication practices with a screen-based simulation, the control group was not given simulation training at this stage of the study, and ended with training on pediatric medication practices, with the training that both groups received in the 2nd step.
Who Masked: Outcomes Assessor
Masking Description: A blind technique was used for the expert who would perform the statistical analysis of the study. The data were tabulated as groups A and B, without using the terms intervention and control group. Statistical analysis of the data was carried out by a statistician other than the person who performed the randomization. The hypotheses of the study were kept confidential in order to prevent the detection bias and risk of bias of the statistician. Thus, internal validity was ensured by randomization and blinding techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Students who agreed to participate in the study and met the inclusion criteria were divided into two groups, intervention and control groups, using a computer-based randomized program. 8 people who did not attend the lecture were not included in the continuation of the study. Randomization occurred among 198 individuals. The intervention group was trained in groups of 10 people with screen-based simulation in the computer laboratory. A pilot study was conducted with the first group. No negative feedback was received. Pilot study group data were also included in the study.
  20 days after the training they received through simulation, the Student Satisfaction and Learning Self-Confidence Scale used in Simulation Training and the Self-Efficacy Scale in Drug Administration in Children were re-administered to Nursing Students. It was applied to both groups through face-to-face interview technique and survey.
  Interventions: Behavioral: screen-based simulation
- control group (No Intervention): The subject of drug administration in children was explained to all participating students using the traditional narrative method.
  Students who agreed to participate in the study and met the inclusion criteria were divided into two groups, intervention and control groups, using a randomized program. Randomization occurred among 198 individuals. The control group was not given training via simulation at this stage of the study and ended with the training that both groups received in step 2.
  Student Satisfaction and Self-Confidence in Learning Scale and Nursing Students Self-Efficacy Scale for Medication Administration in Children were re-administered to both groups and the results were obtained. analyzed. After the data collection process was completed, the control group was also given medication administration training to children through simulation.

INTERVENTIONS:
Behavioral: screen-based simulation — Randomization took place among 198 people. The intervention group was given training on pediatric medication administration through screen-based simulation.
  Arms: intervention group

SUMMARY:
This study was conducted to evaluate the effect of screen-based simulation training on nursing students' self-efficacy in pediatric medication administration and self-confidence in learning.

H1o: Screen-based simulation training has no effect on nursing students' self-efficacy in pediatric medication administration.

H1₁: Education provided with screen-based simulation has an effect on nursing students' self-efficacy in pediatric medication administration.

H2o: Education provided with screen-based simulation has no effect on student satisfaction.

H2₁: Education provided with screen-based simulation has an effect on student satisfaction.

H3o: Education provided with screen-based simulation has no effect on nursing students' self-confidence in learning.

H3₁: Education provided with screen-based simulation has an effect on nursing students' self-confidence in learning.

The lesson was taught to the intervention group using the traditional method. The control group was trained with a screen-based simulation. Self-efficacy and self-confidence in learning results were compared.

DETAILED DESCRIPTION:
This study is an experimental randomized controlled trial conducted to evaluate the effects of screen-based simulation training on nursing students' self-efficacy in pediatric drug administration and their self-confidence in learning.

The population of the study consists of nursing students studying at Balıkesir University Faculty of Health Sciences in the 2023-2024 academic year. There are a total of 206 nursing students in the 2nd and 3rd grades. No sample selection was made in the study, and an attempt was made to reach the population. The study groups were prepared in accordance with the exclusion and inclusion criteria. Two groups were determined as intervention and control groups. The assignment of nursing students to the groups was made by a statistician other than the researcher with a computer-based randomization program in order to prevent bias (https://www.randomizer.org).

The participants were informed about which group they were in as a result of the randomization and were given an appointment to come to the computer laboratory on the specified date and time. Since the researcher managed the study process, researcher blinding could not be performed. The screen-based simulation application of the 10-person subgroups in the intervention group was attempted to be completed as soon as possible within the scope of the computer laboratory appointment and class hours, and interaction between the groups was attempted to be prevented.

A blind technique was used for the expert who would perform the statistical analysis of the study. The data were tabulated as Group A and B without using the terms intervention and control group. The statistical analysis of the data was performed by a statistician other than the person who performed the randomization. The hypotheses of the study were kept confidential in order to prevent the detection bias and risk of bias of the statistician. Thus, internal validity was ensured with the randomization and blinding technique.

The study protocol and reporting of the study were created based on the Consolidated Standards of Reporting Trials (CONSORT), which was specially prepared for randomized controlled studies. Among the 206 people who made up the study group, 8 people who did not attend the theoretical lecture given with the traditional method in the 2nd application step of the study were not included in the study. An intervention and control group were formed from 198 people. There was no person who left the study later or did not want to participate in the study.

The data of the study conducted according to the pre-test-post-test design were collected using the "Sociodemographic Characteristics Form", "Student Satisfaction and Self-Confidence in Learning Scale Used in Simulation Education" and "Children's Medication Self-Efficacy Scale for Nursing Students".

The sociodemographic characteristics form was prepared by the researcher in line with the literature to be applied to the students participating in the study. It consists of a total of 16 items.

It includes questions regarding the demographic information of the students such as gender, age, marital status, high school graduation, and employment status.

Student Satisfaction and Self-Confidence in Learning Scale Used in Simulation Education The validity and reliability of the Turkish form of the "Student Satisfaction and Self-Confidence in Learning Scale" published by the National Nursing Association (NLN) was conducted by Karaçay and Kaya in 2017. Permission was received from Karaçay and Kaya via e-mail for the use of the scale. The scale consists of two sub-dimensions.

These sub-dimensions are:

* Satisfaction in learning
* Self-confidence. The scale is a 5-point Likert type and consists of 13 items in total. The 13th item in the scale is reverse coded. The answer options are 5 = Strongly agree, 4 = Agree, 3 = Undecided: Neither agree nor disagree, 2 = Disagree, 1 = Strongly disagree. Participants are expected to mark the number that best expresses them for each item. The score obtained is obtained by summing the numbers given to the items of the scale. The highest total score that can be obtained from the scale is 65, the lowest score is 13.

A high score that can be obtained from the total of the scale indicates high satisfaction and self-confidence. The internal consistency coefficient of the scale was found to be 0.94.

Self-Efficacy Scale for Nursing Students in Medication Administration in Children

This measurement tool evaluates the self-efficacy of nursing students in preparing and administering medications for pediatric patients. The scale was developed by Bektaş et al. in 2021 and consists of 16 items and two sub-dimensions. Permission was obtained from Bektaş et al. via e-mail for the use of the scale.

These sub-dimensions are designed as;

* Medication preparation sub-dimension for children (items for calculating and obtaining medication dose)
* Medication administration sub-dimension (items for administering the obtained medication).

The expressions of the numbers on the 5-point Likert-type scale are 1=Absolutely inadequate, 2=Somewhat adequate, 3=Partially adequate, 4= Adequate, 5=Absolutely adequate. The lowest score obtained from the scale is 16 and the highest score is 80. The scale has no cut-off point, and as the score increases, the students' self-efficacy in pediatric medication administration increases.

There is no reverse scored item in the scale. Cronbach alpha coefficient was determined as 0.94 for the entire scale, 0.91 for the drug preparation sub-dimension and 0.87 for the drug administration sub-dimension.

All data were recorded and analyzed on the computer using the SPSS (statistical package for social sciences) for Windows 22 program. In the analysis of the data, the assumptions that needed to be met were first tested to decide which tests (parametric/nonparametric tests) would be applied. Kolmogorov-Smirnov, and the kurtosis and skewness values, which are other assumptions of normal distribution, were used to decide on the normality of the distribution.

Mixed design dependent variance analysis was used to examine the difference between dependent variables and the effect of factors on this difference. T-test was applied in dependent groups to determine pre- and post-test score differences, and t-test was applied in independent groups to determine score differences between groups.

A significance level of 0.05 was accepted as the criterion in interpreting whether the obtained values were significant or not.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Volunteering to participate in the research.
* Within the scope of the thesis study, to have attended the theoretical course on drug administration in children given with the traditional lecture method.

Exclusion Criteria:

* Being under 18 years of age,
* Not volunteering to participate in the research,
* Not having attended the theoretical course on drug administration in children, which was given with the traditional lecture method, within the scope of the thesis study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Creation of screen-based simulation | 3 months
  The simulation was prepared in accordance with the good practice standards established by the International Nursing Association for Clinical Simulation and Learning. All animations used in the simulation were taken from the database of the Canva Pro application. The Lumi Education program was used for the software infrastructure. In this way, virtual patients, materials needed while providing care to the patient, necessary information, and process steps were provided to work on interactive screens.
  In the simulation, Voiser voiceover was used to provide education on the subject and to voice the avatar responsible for guiding the student in the simulation.
  A total of 4 scenarios were created. The subject description in the simulation scenarios, patient information (height, weight, disease, etc.), sample dose calculation questions, questions created for virtual patients were created by reviewing the literature, drug administration guide and textbooks.

SECONDARY OUTCOMES:
Data collecting for sociodemographic Characteristics | 2 months
  Sociodemographic characteristics form: It consists of 16 questions including demographic information of students such as gender, age, marital status, high school graduation, employment status.
Data collection for Satisfaction and Self-Confidence | 2 months
  Student Satisfaction and Self-Confidence in Learning Scale Used in Simulation Education: The validity and reliability of the Turkish form of the "Student Satisfaction and Self-Confidence in Learning Scale" published by the National Nursing Association (NLN) was conducted by Karaçay and Kaya in 2017. It has two sub-dimensions as satisfaction in learning and self-confidence. The scale is a 5-point Likert type and consists of 13 items in total. The 13th item in the scale is reverse coded. The highest score that can be obtained from the scale is 65, and the lowest score is 13. A high score that can be obtained from the total scale indicates high satisfaction and self-confidence.30 The internal consistency coefficient of the scale was found to be 0.94. In this study, the Cronbach's Alpha reliability coefficient of the scale was determined as 0.93 for both groups.
Data collecting for Self-Efficacy | 2 months
  Self-Efficacy Scale for Nursing Students in Drug Administration in Children: It evaluates the self-efficacy of nursing students in preparing and administering drugs to child patients. The scale was developed by Bektaş et al. in 2021 and contains 16 items. It consists of two sub-dimensions: drug preparation for children and drug administration. The lowest score obtained from the 5-point Likert-type scale is 16 and the highest score is 80. 31 The Cronbach's alpha coefficient for the entire scale was determined as 0.94. In this study, the Cronbach's Alpha reliability coefficient of the scale was determined as 0.93 for the intervention group and 0.92 for the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Balıkesir University, Balıkesir, Altıeylül, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bayram HC, Ergun S. Effect of screen-based simulation on pediatric drug administration among nursing students: a randomized controlled trial. Rev Esc Enferm USP. 2025 Dec 1;59:e20250249. doi: 10.1590/1980-220X-REEUSP-2025-0249en. eCollection 2025. PMID 41335049